CLINICAL TRIAL: NCT01033799
Title: Effect of the Consumption of a Fermented Milk on Common Infections in Shift-workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU207
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Infectious Diseases; Healthy Subjects; Respiratory Tract Infections; Sore Throat; Sinusitis; Otitis; Bronchitis; Pneumonia; Influenza; Gastroenteritis
Keywords: Probiotic - Lactobacillus casei DN114-001; dairy product - infections - shiftworkers; Common infectious diseases,; occuring in healthy subjects,; including upper respiratory tract infections (defined as rhinopharyngitis, sore throat, sinusitis and otitis),; lower respiratory tract infections (defined as bronchitis,; pneumopathy and flu and flu-like syndromes), and; gastrointestinal tract infection defined as gastroenteritis.
MeSH Terms: conditions — Communicable Diseases; Respiratory Tract Infections; Pharyngitis; Sinusitis; Otitis; Bronchitis; Pneumonia; Influenza, Human; Gastroenteritis; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Product (Sham Comparator)
  Interventions: Other: Non fermented dairy product (control)
- Tested Product (Active Comparator)
  Interventions: Other: Fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel®)

INTERVENTIONS:
Other: Fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel®)
  Arms: Tested Product
Other: Non fermented dairy product (control)
  Arms: Control Product

SUMMARY:
This single-center, randomized, double-blind and controlled study aims to examine the effect of a fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel® = tested product) on the incidence of respiratory and gastro-intestinal common infectious diseases (cumulated number of infections during the intervention period: primary criteria), and on immune functions in healthy shift workers. Volunteers received either 200g/day of tested product (N=500) or control product (N=500) for 3-months, followed by a 1-month follow-up.

ELIGIBILITY:
Inclusion criteria: male and female aged 18-65 years; working in 2- or 3-shift work patterns (including night work); same job position for at least 4.5 months; a 19 to 30 kg/m2 body mass index; no symptoms of CIDs during the 2 weeks before product consumption; agreeing to a written informed consent.

Exclusion criteria: part time work (<90%); allergy/hypersensitivity to components of the study product; severe respiratory allergy; a situation which, in the investigator's opinion, could interfere with optimal participation or constitute a special risk for the volunteer; a history of chronic metabolic/gastro-intestinal disease (except appendectomy); surgery/intervention requiring general anesthesia in the last 4 weeks; administration of systemic/topical treatments likely to interfere with the evaluation parameters in the last 4 weeks; chronic disease requiring antibiotics/antiseptics/anti-inflammatory medications; special medicated diet; chronic/iatrogenic immunodeficiency; cardiac/renal/respiratory insufficiency; severe evolutive/chronic pathology; pregnancy, breast feeding or lacking effective contraception in females; susceptibility not to comply with dietary recommendation during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harrisson Clinical Research Clinical Unit, München, Germany